CLINICAL TRIAL: NCT06724913
Title: Efficacy and Tolerability of a Specialized Food Products for Dietary Therapeutic and Preventive Nutrition Based on Ice Cream (Ice Cream With Brazzein, Maltitol and Oligofructose; Ice Cream With Brazzein, Erythritol, Maltitol and Inulin) Compared to Standard (Sundae) Ice Cream
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology (Other)
Collaborators: Group of companies EFKO (Unknown); Russian Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: OGIG-19-76-30014/2024-1; 19-76-30014-P (Other Grant/Funding Number: Russian Science Foundation)
Record Dates: First submitted 2024-12-06; First posted 2024-12-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Non-Alcoholic Steatohepatitis (NASH); Diabetes Mellitus Type 2 (T2DM)
Keywords: ice cream; NASH; specialized food product; Diabetes mellitus type 2; tolerability; safety; oligofructose; erythritol; inulin; maltitol; blood glycemic monitoring; sundae; brazzein
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2 | interventions — Ice Cream; maltitol; oligofructose; Inulin; Erythritol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Subjects of this arm will receive the following sequence of products: day 1 - ice cream with brazzein, maltitol and oligofructose, day 2 - ice cream with brazzein, erythritol, maltitol and inulin; day 3 - standard ice cream
  Interventions: Other: specialized food product based on ice cream
- Arm 2 (Experimental): Subjects of this arm will receive the following sequence of products: day 1 - ice cream with brazzein, erythritol, maltitol and inulin; day 2 - ice cream with brazzein, maltitol and oligofructose, day 3 - standard ice cream
  Interventions: Other: specialized food product based on ice cream 2
- Arm 3 (Experimental): Subjects of this arm will receive the following sequence of products: day 1 - standard ice cream; day 2 - ice cream with brazzein, maltitol and oligofructose, day 3 - ice cream with brazzein, erythritol, maltitol and inulin
  Interventions: Other: specialized food product based on ice cream 3

INTERVENTIONS:
Other: specialized food product based on ice cream — Day 1: ice cream with 0.014% brazzein, 6% maltitol and 8% oligofructose Day 2: ice cream with 0.014% brazzein, 7.5% erythritol, 2.5% maltitol and 4% inulin Day 3: standard ice cream (12% fat)
  Other Names: ice cream with brazzein, maltitol and oligofructose; ice cream with brazzein, maltitol, inulin, erythritol; standard ice cream (sundae)
  Arms: Arm 1
Other: specialized food product based on ice cream 2 — Day 1: ice cream with 0.014% brazzein, 7.5% erythritol, 2.5% maltitol and 4% inulin Day 2: ice cream with 0.014% brazzein, 6% maltitol and 8% oligofructose Day 3: standard ice cream (12% fat)
  Arms: Arm 2
Other: specialized food product based on ice cream 3 — Day 1: standard ice cream (12% fat) Day 2: ice cream with 0.014% brazzein, 6% maltitol and 8% oligofructose Day 3: ice cream with 0.014% brazzein, 7.5% erythritol, 2.5% maltitol and 4% inulin
  Arms: Arm 3

SUMMARY:
This is a double-blind, randomized, comparative controlled cross-over study of efficacy and tolerability of 2 specialized food products based on ice cream compared to the standard (sundae) ice cream for patients with non-alcoholic fatty liver disease with or without type 2 diabetes mellitus. On 3 consecutive days eligible subjects will receive a portion of specialized food products with breakfast (ice cream with brazzein, maltitol and oligofructose; ice cream with brazzein, erythritol, maltitol and inulin; standard ice cream (sundae)) followed by the standard ration. Tolerability will be assessed based on specialized scales and formal questioning. Glucose monitoring will be performed with the use of prolonged blood glucose monitoring system (FreeStyle Libre 2, Abbott Diabetes Care, USA)

DETAILED DESCRIPTION:
An organoleptic evaluation study phase preceded the main active intervention phase of the study. During this phase, all three types of ice cream were evaluated using a 5-point hedonic scale (1 = dislike extremely, 3 = neither like nor dislike, 5 = like extremely) for overall impression, flavor, color, appearance, aroma, and texture. Portions of 100 g of the ice cream were used with proper labelling (three-digit code) for randomization and supporting crossover design. The evaluation was performed as one portion per day and organized due to technical reasons as two round evaluations, in which one round included standard ice cream and the 1st special product, and the second round included standard ice cream and the 2nd special product. There were 3 days washout period between rounds to prevent carryover effects between the tested products. The percentage of ice cream consumed was determined by weighing the remaining portion of each ice cream after testing.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate based on signed written informed consent;
* controlled glycemia. If stable glycemia is achieved on treatment, the following requirements should be met:
* no qualitative changes in treatment within 6 months before enrollment (i.e., the introduction of a new antidiabetic therapy);
* doses of anti-diabetic medications should be stable for 6 month in patients who receive metformin, gliptins, sulfonylureas, sodium/glucose cotransporter 2 (SGLT-2) inhibitors, glucagon-like peptide 1 agonists (GLP-1) or insulin.
* no new medications during participation in the study

Exclusion Criteria:

* Pregnancy and breastfeeding;
* Liver cirrhosis based on liver histology, or liver stiffness measurement (LSM > or = 14 kPa by Fibroscan), or APRI > or= 1; or BARD score > or = 2.
* Chronic heart failure (I-IV class by NYHA).
* Past bariatric surgery.
* Clinically relevant acute cardiovascular event within 6 months prior to screening.
* Uncontrolled arterial hypertension despite optimal antihypertensive therapy.
* Diabetes mellitus type 1.
* The level of glycated hemoglobin [HbA1c] >9.0%.
* Hypersensitivity to the studied product or any of its components.
* The intake of any medications that may affect the absorption, distribution, metabolism or excretion of investigational products or may lead to the induction or inhibition of microsomal enzymes (for example, indomethacin) - from the moment of randomization to the end of treatment.
* Any medical conditions that may significantly affect life expectancy, including known cancers;
* Any clinically significant immunological, endocrine, hematological, gastrointestinal, neurological, tumor or psychiatric diseases;
* Mental instability or incapacity, which may impact the ability to give informed consent, take part in the study, or affect the ability to comply with the requirements of the study protocol.
* Positive HIV blood antigen test.
* Serum aspartate aminotransferase (AST) and/or ALT >10 x upper normal limits.
* conjugated bilirubin > 26 mcmol/l due to changes in liver function (patients with Gilbert's disease are allowed to the study).

  * The international normalized ratio is >1.40 due to changes in liver function.
  * Platelet count <100 x 10^9/L due to portal hypertension.
  * Clinically significant renal dysfunction, including nephrotic syndrome, chronic kidney disease (determined based on the estimated glomerular filtration rate [eGFR] less than 60 ml/min/1.73 m^2).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
mean daily glucose change | baseline and day 1
  mean blood glucose concentration based on monitoring system
mean daily glucose change | baseline and day 2
  Mean daily blood glucose concentrations based on monitoring system
mean daily glucose change | baseline and day 3
  Mean daily blood glucose concentrations based on monitoring system
mean daily glucose change | baseline and day 4
  Mean daily blood glucose concentrations based on monitoring system
stool frequency | baseline and day 1
  stool frequency (formal)
stool frequency | baseline and day 2
  stool frequency (formal)
stool frequency | baseline and day 3
  stool frequency (formal)
stool frequency | baseline and day 4
  stool frequency (formal)
stool form | baseline and day 1
  stool form according to Bristol stool scale
stool form | baseline and day 2
  stool form according to Bristol stool scale
stool form | baseline and day 3
  stool form according to Bristol stool scale
stool form | baseline and day 4
  stool form according to Bristol stool scale

OTHER OUTCOMES:
product organoleptic assessment | An organoleptic evaluation study phase
  5-point hedonic scale (1 = dislike extremely, 3 = neither like nor dislike, 5 = like extremely) for overall impression, flavor, color, appearance, aroma, and texture

CONTACTS AND LOCATIONS:
Overall Officials: Vasily Isakov, MD, PhD, Professor, Study Chair — Department of Gastroenterology, Hepatology and Nutrition. Federal Research Centre of Nutrition, Biotechnology and Food Safety, Moscow, Russia
Locations (1):
- Dpt Gastroenterology, Hepatology and Nutrition, Federal Research Centre of Nutrition and Biotechnology, Kashirskoye shosse, bld 21, Moscow, Russia., Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
Depersonalized study data will be available upon reasonable request to principal investigator
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 5 years after study completion